CLINICAL TRIAL: NCT07199621
Title: Comparing Scissors Versus Scalpel in Uterine Incision During Cesarean Section
Brief Title: Comparing Bet Scissors &Scalpel in Uterotomy in CS
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nayra Hussien Ahmed, Doctor, Assiut University
Other Study IDs: uterotomy by scissor & scalpel
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Blood Loss in Uterotomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: uterine incision by scissors versus scalpel — procedure in uterotomy in cs

SUMMARY:
To compare between rate of blood loss in uterine incision using scissors and scalpel in caesarean section

DETAILED DESCRIPTION:
In present-day obstetrics, cesarean delivery occurs in one in three women in the United States, and in up to four of five women in some regions of the world . . Concurrently, despite attempts to encourage vaginal birth after previous cesareans, the cesarean delivery rate increased steadily from 5 to 30-32% over the last 10 years, with a parallel increase in costs as well as short- and long-term maternal, neonatal and childhood complications( 1). Approximately 30% of women will experience a maternal or neonatal complication during childbirth. Both cesarean and vaginal delivery is associated with well-known measurable short- and long-term maternal and neonatal complications and benefits.(2 ) the most concerning complications from cesareans are the neonatal respiratory morbidity and the impact on a mother's future reproductive health, including the risk of abnormal placentation such as placenta previa or accreta.( 3) Fetal laceration injury at cesarean delivery is not rare, especially when it is performed for nonvertex presentation. The minority of obstetric records show documentation of such lacerations, suggesting that this complication often may not be recognized by obstetricians 4. During urgent CS, the surgeon should bear in mind that the presence of PROM or meconium-stained amniotic fluid should prompt extra care and application of preventive measures to decrease blood loss .(.4) To the best of our knowledge, no studies have investigated the association of type of uterotomy and incidence of accidental fetal lacerations. For this reason, in this study we evaluated whether using scissors instead of scalpel in uterotomy can prevent maternal blood loss at time of CS (.5)

ELIGIBILITY:
Inclusion Criteria:

* 1.pregnant women age 18-40 years 2.Gestational age between 37-42 weeks 3.Admitted for Elective caesarean delivery in the hospital

Exclusion Criteria:

* 1.placental pervia and accreta 2.cases refused to be recruited in the study 3. obstructed labor

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: pregnant women age 18-40 years ,their gestational age between 37-42 weeks admitted for Elective CS
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Comparing between Maternal blood loss in uterotomy using by scissors and scalpel | baseline

REFERENCES:
- [Background] Har-Shai L, Kreichman R, Kedar R, Osovsky M, Chen R, Lavi I, Metanes I, Segal M, Ofek SE, Mattar S, Hassan S, Kramer A, Bryzgalin L, Ad-El D, Sagi-Dain L, Lavie O, Har-Shai Y. Risk factors associated with accidental fetal skin lacerations during cesarean delivery. Int J Gynaecol Obstet. 2023 Jan;160(1):131-135. doi: 10.1002/ijgo.14273. Epub 2022 Jun 2. PMID 35598118
- [Background] Smith JF, Hernandez C, Wax JR. Fetal laceration injury at cesarean delivery. Obstet Gynecol. 1997 Sep;90(3):344-6. doi: 10.1016/s0029-7844(97)00284-6. PMID 9277641
- [Background] Lee YM, D'Alton ME. Cesarean delivery on maternal request: maternal and neonatal complications. Curr Opin Obstet Gynecol. 2008 Dec;20(6):597-601. doi: 10.1097/GCO.0b013e328317a293. PMID 18989137
- [Background] Gregory KD, Jackson S, Korst L, Fridman M. Cesarean versus vaginal delivery: whose risks? Whose benefits? Am J Perinatol. 2012 Jan;29(1):7-18. doi: 10.1055/s-0031-1285829. Epub 2011 Aug 10. PMID 21833896
- [Background] Antoine C, Young BK. Cesarean section one hundred years 1920-2020: the Good, the Bad and the Ugly. J Perinat Med. 2020 Sep 4;49(1):5-16. doi: 10.1515/jpm-2020-0305. PMID 32887190